CLINICAL TRIAL: NCT00864383
Title: A Randomised Placebo - Controlled Double Blind Trial Comparing 1) a Two Month Intensive Phase of Ethambutol, Moxifloxacin, Rifampicin, Pyrazinamide Versus the Standard Regimen (Ethambutol, Isoniazid, Rifampicin, Pyrazinamide) and 2) a Treatment Shortening Regimen Comparing Two Months Moxifloxacin, Isoniazid, Rifampicin, Pyrazinamide Followed by Two Months Moxifloxacin, Isoniazid, Rifampicin Versus the Standard Regimen (Two Months Ethambutol, Isoniazid, Rifampicin, Pyrazinamide Followed by Four Months Isoniazid and Rifampicin) for the Treatment of Adults With Pulmonary Tuberculosis
Brief Title: Controlled Comparison of Two Moxifloxacin Containing Treatment Shortening Regimens in Pulmonary Tuberculosis
Acronym: REMoxTB
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Global Alliance for TB Drug Development (Other)
Collaborators: European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government); University College, London (Other); Bayer Healthcare Pharmaceuticals, Inc./Bayer Schering Pharma (Industry); Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REMoxTB; ISRCTN85595810
Record Dates: First submitted 2009-03-17; First posted 2009-03-18 (Estimated); Results first posted 2015-05-25 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-02

CONDITIONS: Pulmonary Tuberculosis
MeSH Terms: conditions — Tuberculosis, Pulmonary | interventions — Moxifloxacin; Ethambutol; Isoniazid; Pyrazinamide; Rifampin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Regimen 1 - 2EHRZ/4HR (control regimen) (Placebo Comparator): * Eight weeks of chemotherapy with Ethambutol, Isoniazid, Rifampicin and Pyrazinamide plus the Moxifloxacin placebo, followed by
  * Nine weeks of Isoniazid and Rifampicin plus the Moxifloxacin placebo, followed by
  * Nine weeks of Isoniazid and Rifampicin only.
  Interventions: Drug: Moxifloxacin, Ethambutol, Isoniazid, Pyrazinamide & Rifampicin
- Regimen 2 - 2MHRZ/2MHR (Experimental): * Eight weeks of chemotherapy with Moxifloxacin, Isoniazid, Rifampicin and Pyrazinamide plus the Ethambutol placebo, followed by
  * Nine weeks of Moxifloxacin, Isoniazid and Rifampicin, followed by
  * Nine weeks of the Isoniazid placebo and the Rifampicin placebo.
  Interventions: Drug: Moxifloxacin, Ethambutol, Isoniazid, Pyrazinamide & Rifampicin
- Regimen 3 - 2EMRZ/2MR (Experimental): * Eight weeks of chemotherapy with Ethambutol, Moxifloxacin, Rifampicin and Pyrazinamide plus the Isoniazid placebo, followed by
  * Nine weeks of Moxifloxacin and Rifampicin plus the Isoniazid placebo, followed by
  * Nine weeks of the Isoniazid placebo and the Rifampicin placebo
  Interventions: Drug: Moxifloxacin, Ethambutol, Isoniazid, Pyrazinamide & Rifampicin

INTERVENTIONS:
Drug: Moxifloxacin, Ethambutol, Isoniazid, Pyrazinamide & Rifampicin — Moxifloxacin 400 mg Rifampicin < 45 kg 450 mg > 45 kg 600 mg Isoniazid 300 mg Pyrazinamide < 40 kg 25 mg/kg rounded to nearest 500 mg* 40-55 kg 1000 mg > 55 kg - 75 kg 1500 mg > 75 kg 2000 mg Ethambutol < 40 kg 15 mg/kg rounded to nearest 100 mg 40-55 kg 800 mg > 55 kg - 75 kg 1200 mg > 75 kg 1600 mg *For pyrazinamide dosing in patients < 40 kg, 1000 mg used instead of 500 mg
  All treatment is taken daily, for a duration of up to 26 weeks depending on treatment arm.
  Other Names: Avelox; Avelon; Avalox; Myambutol; Nydrazid; Rifampin; Rifadin

SUMMARY:
REMoxTB is a study for the "Rapid Evaluation of Moxifloxacin in the treatment of sputum smear positive tuberculosis". REMoxTB aims to find and evaluate new drugs and regimens that shorten the duration of tuberculosis therapy.

The purpose of REMoxTB is to evaluate the efficacy, safety and acceptability of two moxifloxacin-containing treatment combinations to determine whether substituting ethambutol with moxifloxacin in one combination, and/or substituting isoniazid with moxifloxacin in another combination, makes it possible to reduce the duration of treatment for TB.

DETAILED DESCRIPTION:
The current recommended treatments for tuberculosis (TB) require a patient to take multiple drugs for six to eight months. Because the course of therapy is long, many patients do not adhere to treatment and as a consequence they have a poor outcome. In these cases either the sputum is not cleared of the bacteria causing tuberculosis, or the disease returns again (called relapse). Response to medication can be monitored during treatment by collecting regular sputum samples and examining these samples by culture, for the organisms that cause tuberculosis.

The commonly used drugs to treat tuberculosis are rifampicin, isoniazid, ethambutol and pyrazinamide. Previous studies in animals and in humans suggest that a new drug called moxifloxacin may also be an effective treatment in tuberculosis. Moreover, promising laboratory studies on mice suggest that moxifloxacin may enable the total duration of chemotherapy to be reduced to four months, which would be a significant improvement for patients taking medication for tuberculosis.

This study will involve comparisons that are designed to assess whether substituting moxifloxacin for individual drugs in existing treatment combinations will enable tuberculosis treatment to be shortened. Patients selected for the study will be allocated to one of three treatment groups. The first group will be given six months standard treatment. A second group will receive moxifloxacin substituted for ethambutol, as part of a four month regimen, to see whether the shorter treatment is not inferior to the standard six month treatment. The third group will receive moxifloxacin substituted for isoniazid, as part of a four month regimen, to see whether the shorter treatment is not inferior to the standard six month treatment.

Hypotheses:

1. In treatment-naïve adults with active pulmonary TB treated with eight weeks of moxifloxacin (M), isoniazid (H), rifampicin (R) and pyrazinamide (Z) (i.e. a standard regimen where moxifloxacin is substituted for ethambutol (E)), followed by nine weeks of moxifloxacin, isoniazid and rifampicin, followed by nine weeks of placebo, the proportion of patients who experience treatment failure or disease relapse in the twelve months following treatment completion will not be inferior to that observed in patients who are treated with a standard regimen (eight weeks of ethambutol, isoniazid, rifampicin and pyrazinamide followed by eighteen weeks of isoniazid plus rifampicin) (Comparison 1).
2. In treatment-naïve adults with active pulmonary TB treated with eight weeks of ethambutol, moxifloxacin, rifampicin and pyrazinamide (i.e. a standard regimen where moxifloxacin is substituted for isoniazid), followed by nine weeks of moxifloxacin and rifampicin followed by nine weeks of placebo, the proportion of patients who experience treatment failure or disease relapse in the twelve months following treatment completion will not be inferior to that observed in patients who are treated with a standard regimen (eight weeks of ethambutol, isoniazid, rifampicin and pyrazinamide followed by eighteen weeks of isoniazid plus rifampicin) (Comparison 2).

ELIGIBILITY:
Inclusion Criteria:

* Signed written consent or witnessed oral consent in the case of illiteracy, before undertaking any trial related activity.
* Two sputum specimens positive for tubercle bacilli on smear microscopy at least one of which must be processed and positive at the study laboratory.
* Aged 18 years or over.
* No previous anti-tuberculosis chemotherapy.
* A firm home address that is readily accessible for visiting and willingness to inform the study team of any change of address during the treatment and follow-up period.
* Agreement to participate in the study and to give a sample of blood for HIV testing (see appendices 1 & 2).
* Pre-menopausal women must be using a barrier form of contraception or be surgically sterilised or have an IUCD in place.
* Laboratory parameters performed up to 14 days before enrolment.

  * Serum aspartate transaminase (AST) and alanine transaminase (ALT) activity less than 3 times the upper limit of normal.
  * Serum total bilirubin level less than 2.5 times upper limit of normal. Creatinine clearance (CrCl) level greater than 30 mls/min.
  * Haemoglobin level of at least 7.0 g/dL.
  * Platelet count of at least 50x109cells/L.
  * Serum potassium greater than 3.5 mmol/L.
* Negative pregnancy test (women of childbearing potential).

Exclusion Criteria:

* Unable to take oral medication.
* Previously enrolled in this study.
* Received any investigational drug in the past 3 months.
* Received an antibiotic active against M. tuberculosis in the last 14 days (fluoroquinolones, macrolides, standard anti-tuberculosis drugs).
* Any condition that may prove fatal during the first two months of the study period.
* TB meningitis or other forms of severe tuberculosis with high risk of a poor outcome
* Pre-existing non-tuberculosis disease e.g. diabetes, liver or kidney disease, blood disorders,peripheral neuritis, chronic diarrhoeal disease in which the current clinical condition of the patient is likely to prejudice the response to, or assessment of treatment.
* Pregnant or breast feeding.
* Suffering from a condition likely to lead to uncooperative behaviour e.g. psychiatric illness or alcoholism.
* Contraindications to any medications in the study regimens.
* Known to have congenital or sporadic syndromes of QTc prolongation or receiving concomitant medication reported to increase the QTc interval (e.g. amiodarone, sotalol, disopyramide, quinidine, procainamide, terfenadine).
* Known allergy to any fluoroquinolone antibiotic or history of tendinopathy associated with quinolones.
* Patients already receiving anti-retroviral therapy.
* Patients whose initial isolate is shown to be multiple drug resistant (i.e. resistant to rifampicin and isoniazid) or monoresistant to rifampicin, or resistant to any fluoroquinolone)
* Weight less than 35kg
* HIV infection with CD4 count less than 250 cells/µL.
* End stage liver failure (class Child-Pugh C).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1931 (Actual)
Dates: Start 2008-01; Primary Completion 2013-10 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen H Gillespie, MB BCh BAO MD DSc, Study Director — University of St Andrews; Andrew Nunn, BSc MSc, Principal Investigator — MRC Clinical Trials Unit; Sarah K Meredith, MB BS MSc, Principal Investigator — MRC Clinical Trials Unit; Timothy D McHugh, BSc PhD CSi, Principal Investigator — Centre for Medical Microbiology, Royal Free and University College Medical School; Ali Zumla, BSc MBChB MSc PhD, Principal Investigator — Centre for International Health, Royal Free and University College Medical School; Alexander Pym, MB BMRCP PhD, Principal Investigator — Unit for Clinical & Biomedical TB Research, MRC Durban; Peter Mwaba, MB ChB MMed PhD, Principal Investigator — University Teaching Hospital; Noel Sam, MMed MD, Principal Investigator — Kilimanjaro Christian Medical Centre; Andreas Diacon, BM MD, Principal Investigator — Tiervlei Trial Center and University of Stellenbosch; Rodney Dawson, MB ChB FCP, Principal Investigator — Centre for TB Research and Innovation, UCT Lung Institute; Evans Amukoye, MBChB. Mmed (Paediatric), Principal Investigator — Centre for Respiratory Disease Research at KEMRI; Leonard Maboko, MD MSc PhD, Principal Investigator — NIMR - Mbeya Medical Research Programme; Ian Sanne, MBBCH FCP(SA), Principal Investigator — Clinical HIV Research Unit (CHRU), Westdene; Cheryl Louw, MBChB, Principal Investigator — Madibeng Centre For Research, Brits; Mengqui Gao, MD, Principal Investigator — Beijing Tuberculosis and Thoracic Tumor Research Institute; Qing Zhang, MD, Principal Investigator — Shanghai Pulmonary Hospital, Shanghai, China; Xiexiu Wang, MD, Principal Investigator — TB Institute, Tianjin; Aziah Mahayiddin, MD, Principal Investigator — Institute of Respiratory Medicine (IPR) Jalan Pahang, Malaysia; Watchara Boonsawat, MD PhD, Principal Investigator — Srinagarind Hospital, Division of Pulmonary Medicine, Khon Kaen University; Charoen Chuchottaworn, MD, Principal Investigator — Chest Disease Institute (CDI), Ministry of Public Health, Nonthaburi; Pairaj Kateruttanakul, MD, Principal Investigator — Rajavithi Hospital, Division of Pulmonary, Department of Medicine, Bangkok; Gerardo Amaya-Tapia, MD, Principal Investigator — Hospital General de occidente de la secretaria, Seattle, Mexico; Stephen Murray, M.D, PhD, Principal Investigator — Global Alliance for TB Drug Development; Michael Brown, BA, BM, BCh, MRCP, PhD, DTM&H, Principal Investigator — London School of Hygiene and Tropical Medicine; Rakesh Lal, MD, Principal Investigator — Centre for Advanced Lung and Sleep Disorders, New Delhi, India; Rakesh Mittal, MBBS MD, Principal Investigator — Dr. Mittal's Clinic, Balaji Medical Store, New Delhi, India; A K Jain, MBBS FICA, Principal Investigator — Diligent Hospital, New Delhi, India; Mahesh Kapoor, MBBS DTCD, Principal Investigator — A One Hospital, New Delhi, India; D K Chauhan, MBBS, Principal Investigator — Dr D.K. Chauhan, New Delhi, India; Mahip Saluja, M.D, Principal Investigator — Dr. Mahip Saluja Clinic, Meerut, U.P. India; Neeraj Gupta, MD, Principal Investigator — Dr. Neeraj Gupta, Firozabad ,U.P, India; Subodh Katiyar, MD, Principal Investigator — Dr Subodh, Swaroop Nagar,Kanpur, India; Nirmal K Jain, MD, Principal Investigator — Dr.Nirmal Kumar Jain, Jaipur, India; Komal Gupta, M.D, Principal Investigator — Kilkari , Lucknow , India; Fahad Khan, MD, Principal Investigator — New City Hospital and Trauma Centre, Lucknow, India; Vaibhav Gupta, MD, Principal Investigator — Saanvi MultiSpeciality Clinic, Moradabad, UP, India,; Suraj P Sondhi, MD, Principal Investigator — Dr. S. P. Sondhi Clinic , Meerut U.P India; Siddharth Agarwal, MD, Principal Investigator — Siddharth Nursing Home, Agra, U.P India; Sanjay Teotia, M.D, Principal Investigator — Dr. Sanjay Teotia Clinic, Meerut, U.P , India; S PS Chauhan, MD, Principal Investigator — Dr. SPS Chauhan, Firozabad, U.P-India,; Mahesh Mishra, MD, Principal Investigator — Mahatma Gandhi Medical College& Hospital , Jaipur, India; Ashish Rohatgi, DTCD, Principal Investigator — Ish Medical Centre and Respiratory Lab, New Delhi- India; Om P Rai, MD, Principal Investigator — Guru Tej Bahadur Hospital, Kanpur India; Pawan Varshneya, MD, Principal Investigator — Varshneya Chest Clinic & Eye Care Centre, Aligarh, UP India; R K Garg, MD, Principal Investigator — Dr. R. K. Garg's Clinic, U.P, India; Vinod K Karhana, M.D, Principal Investigator — Prakash Devi Memorial Medical Centre,New Delhi, India; Vijay K Khurana, M.D, Principal Investigator — Ram-Tej Hospital, Agra, India; Surya Kant, MD, FCCP, FNCP, FCAI, Principal Investigator — Dr.Surya Kant, Lucknow, India; Shalini Arya, MD, Principal Investigator — Arya Chest Clinic, Meerut, UP,India; Ashok K Singh, MD, FCCP, FCCS, Principal Investigator — Pulmonary Care and Sleep Clinic, Kanpur, India; Bhanu P Singh, MD, FCCP, Principal Investigator — Surya Chest Foundation, Lucknow India; Chandra P Singh, MD, Principal Investigator — Jigyasa Medical Center,Uttar Pradesh, India; Arun Aggarwal, MD, Principal Investigator — Indra Nursing Home and Maternity Centre, Uttar Pradesh, India; Anjula Bhargava, MS, Principal Investigator — Rajul Nursing Home, Sasni Gate, Aligarh, UP India; Angela Crook, Principal Investigator — MRC Clinical Trials Unit; Salome Charalambous, Principal Investigator — The Aurum Institute, Tembisa Hospital, South Africa; Lerato Mohapi, Principal Investigator — Soweto Perinatal HIV Research Unit, Johannesburg, South Africa; Nesri Padayatchi, Principal Investigator — Caprisa eThakwini Research Facility, Durban, South Africa; Sandy Pillay, Principal Investigator — International Clinical Trials Unit, Durban, South Africa
Locations (47):
- China (3):
  - Beijing Tuberculosis and Thoracic Tumor Research Institute, Beijing
  - Shanghai Pulmonary Hospital, Shanghai
  - TB Institute, Tianjin
- India (30):
  - Nirmal Kumar Jain, Jaipur, Rajasthan
  - Mahatma Gandhi Medical College& Hospital, Jaipur, Rajsthan
  - Ram-Tej Hospital,, Agra, Uttar Pradesh
  - Siddharth Nursing Home,, Agra, Uttar Pradesh
  - Rajul Nursing Home, Aligarh, Uttar Pradesh
  - Varshneya Chest Clinic & Eye Care Centre, Aligarh, Uttar Pradesh
  - Dr. Neeraj Gupta Clinic, Firozabad, Uttar Pradesh
  - S.P.S Chauhan Clinic, Firozabad, Uttar Pradesh
  - Dr. R. K. Garg's Clinic,, Ghaziabad, Uttar Pradesh
  - Indra Nursing Home and Maternity Centre, Ghaziabad, Uttar Pradesh
  - Dr. AK Singh Clinic, Kanpur, Uttar Pradesh
  - Dr. S. K. Katiyar, Swaroop Nagar,, Kanpur, Uttar Pradesh
  - Guru Tej Bahadur Hospital, Kanpur, Uttar Pradesh
  - Dr. Komal Gupta, Lucknow, Uttar Pradesh
  - New City Hospital and Trauma Centre,, Lucknow, Uttar Pradesh
  - Surya Chest Foundation,, Lucknow, Uttar Pradesh
  - Surya Kant Clinic, Lucknow, Uttar Pradesh
  - Arya Chest Clinic, UP,India, Meerut, Uttar Pradesh
  - Dr. Mahip Saluja Clinic, U.P., Meerut, Uttar Pradesh
  - Dr. S. P. Sondhi Clinic,, Meerut, Uttar Pradesh
  - Sri Ram Plaza, Meerut, Uttar Pradesh
  - Jigyasa Medical Center, Morādābād, Uttar Pradesh
  - Saanvi MultiSpeciality Clinic,, Morādābād, Uttar Pradesh
  - A-One Hospital, Delhi
  - Dr. D.K. Chauhan, New Delhi
  - Centre for advanced lung and sleep disorders, New Delhi
  - Dr. Mittal's clinic, New Delhi
  - Diligent Hospital, New Delhi
  - Ish Medical Centre and Respiratory Lab,, New Delhi
  - Smt Prakash Devi Memorial Medical Centre,, New Delhi
- Centre for Respiratory Disease Research at KEMRI, Nairobi, Kenya
- Institute of Respiratory Medicine (IPR) Jalan Pahang, Kuala Lumpur, Malaysia
- Hospital General de Occidente de la secretaria, Guadalajara, Seattle, Mexico
- South Africa (5):
  - Madibeng centre for Research, 40 Pienaar Street,, Madibeng, Brits
  - Clinical HIV Research Unit (CHRU), Johannesburg, Westdene
  - Centre for TB Research and Innovation, University of Cape Town Lung Institute, Cape Town
  - Tiervlei Trial Center and University of Stellenbosch, Cape Town
  - Unit for Clinical & Biomedical TB Research, MRC Durban, Durban
- Tanzania (2):
  - NIMR Mbeya Medical Research Programme, Mbeya
  - Kilimanjaro Christian Medical Centre, Moshi
- Thailand (3):
  - Srinagarind Hospital, Division of Pulmonary Medicine, Khon Kaen University, Khon Kaen, Mueang
  - Chest Disease Institute (CDI), Ministry of Public,, Nonthaburi, Mueang
  - Rajavithi Hospital, Division Of Pulmonary Medicine, Bangkok, Phayathai
- University Teaching Hospital, Lusaka, Zambia

REFERENCES:
- [Background] Bryant JM, Harris SR, Parkhill J, Dawson R, Diacon AH, van Helden P, Pym A, Mahayiddin AA, Chuchottaworn C, Sanne IM, Louw C, Boeree MJ, Hoelscher M, McHugh TD, Bateson AL, Hunt RD, Mwaigwisya S, Wright L, Gillespie SH, Bentley SD. Whole-genome sequencing to establish relapse or re-infection with Mycobacterium tuberculosis: a retrospective observational study. Lancet Respir Med. 2013 Dec;1(10):786-92. doi: 10.1016/S2213-2600(13)70231-5. Epub 2013 Nov 21. PMID 24461758
- [Background] Friedrich SO, Rachow A, Saathoff E, Singh K, Mangu CD, Dawson R, Phillips PP, Venter A, Bateson A, Boehme CC, Heinrich N, Hunt RD, Boeree MJ, Zumla A, McHugh TD, Gillespie SH, Diacon AH, Hoelscher M; Pan African Consortium for the Evaluation of Anti-tuberculosis Antibiotics (PanACEA). Assessment of the sensitivity and specificity of Xpert MTB/RIF assay as an early sputum biomarker of response to tuberculosis treatment. Lancet Respir Med. 2013 Aug;1(6):462-70. doi: 10.1016/S2213-2600(13)70119-X. Epub 2013 Jul 1. PMID 24429244
- [Result] Gillespie SH, Crook AM, McHugh TD, Mendel CM, Meredith SK, Murray SR, Pappas F, Phillips PP, Nunn AJ; REMoxTB Consortium. Four-month moxifloxacin-based regimens for drug-sensitive tuberculosis. N Engl J Med. 2014 Oct 23;371(17):1577-87. doi: 10.1056/NEJMoa1407426. Epub 2014 Sep 7. PMID 25196020
- [Derived] Weir IR, Dufault SM, Phillips PPJ. Estimands for clinical endpoints in tuberculosis treatment randomized controlled trials: a retrospective application in a completed trial. Trials. 2024 Mar 12;25(1):180. doi: 10.1186/s13063-024-07999-w. PMID 38468320
- [Derived] Weir IR, Dufault SM, Phillips PP. Estimands for clinical endpoints in Tuberculosis treatment randomized controlled trials: a retrospective application in a completed trial. Res Sq [Preprint]. 2023 Nov 9:rs.3.rs-3486707. doi: 10.21203/rs.3.rs-3486707/v1. PMID 37986887
- [Derived] Rachow A, Saathoff E, Mtafya B, Mapamba D, Mangu C, Rojas-Ponce G, Ntinginya NE, Boeree M, Heinrich N, Gillespie SH, Hoelscher M; PanACEA-Consortium. The impact of repeated NALC/NaOH- decontamination on the performance of Xpert MTB/RIF assay. Tuberculosis (Edinb). 2018 May;110:56-58. doi: 10.1016/j.tube.2018.04.001. Epub 2018 Apr 5. PMID 29779774
- [Derived] Phillips PP, Mendel CM, Burger DA, Crook AM, Nunn AJ, Dawson R, Diacon AH, Gillespie SH. Limited role of culture conversion for decision-making in individual patient care and for advancing novel regimens to confirmatory clinical trials. BMC Med. 2016 Feb 4;14:19. doi: 10.1186/s12916-016-0565-y. PMID 26847437

RESULTS

PARTICIPANT FLOW:
Groups:
- Regimen 1 - 2EHRZ/4HR (Control Regimen): * Eight weeks of chemotherapy with Ethambutol, Isoniazid, Rifampicin and Pyrazinamide plus the Moxifloxacin placebo, followed by
  * Nine weeks of Isoniazid and Rifampicin plus the Moxifloxacin placebo, followed by
  * Nine weeks of Isoniazid and Rifampicin only.
  Moxifloxacin, Ethambutol, Isoniazid, Pyrazinamide & Rifampicin: Moxifloxacin 400 mg Rifampicin < 45 kg 450 mg > 45 kg 600 mg Isoniazid 300 mg Pyrazinamide < 40 kg 25 mg/kg rounded to nearest 500 mg* 40-55 kg 1000 mg > 55 kg - 75 kg 1500 mg > 75 kg 2000 mg Ethambutol < 40 kg 15 mg/kg rounded to nearest 100 mg 40-55 kg 800 mg > 55 kg - 75 kg 1200 mg > 75 kg 1600 mg *For pyrazinamide dosing in patients < 40 kg, 1000 mg used instead of 500 mg
  All treatment is taken daily, for a duration of up to 26 weeks depending on treatment arm.
- Regimen 2 - 2MHRZ/2MHR: * Eight weeks of chemotherapy with Moxifloxacin, Isoniazid, Rifampicin and Pyrazinamide plus the Ethambutol placebo, followed by
  * Nine weeks of Moxifloxacin, Isoniazid and Rifampicin, followed by
  * Nine weeks of the Isoniazid placebo and the Rifampicin placebo.
  Moxifloxacin, Ethambutol, Isoniazid, Pyrazinamide & Rifampicin: Moxifloxacin 400 mg Rifampicin < 45 kg 450 mg > 45 kg 600 mg Isoniazid 300 mg Pyrazinamide < 40 kg 25 mg/kg rounded to nearest 500 mg* 40-55 kg 1000 mg > 55 kg - 75 kg 1500 mg > 75 kg 2000 mg Ethambutol < 40 kg 15 mg/kg rounded to nearest 100 mg 40-55 kg 800 mg > 55 kg - 75 kg 1200 mg > 75 kg 1600 mg *For pyrazinamide dosing in patients < 40 kg, 1000 mg used instead of 500 mg
  All treatment is taken daily, for a duration of up to 26 weeks depending on treatment arm.
- Regimen 3 - 2EMRZ/2MR: * Eight weeks of chemotherapy with Ethambutol, Moxifloxacin, Rifampicin and Pyrazinamide plus the Isoniazid placebo, followed by
  * Nine weeks of Moxifloxacin and Rifampicin plus the Isoniazid placebo, followed by
  * Nine weeks of the Isoniazid placebo and the Rifampicin placebo
  Moxifloxacin, Ethambutol, Isoniazid, Pyrazinamide & Rifampicin: Moxifloxacin 400 mg Rifampicin < 45 kg 450 mg > 45 kg 600 mg Isoniazid 300 mg Pyrazinamide < 40 kg 25 mg/kg rounded to nearest 500 mg* 40-55 kg 1000 mg > 55 kg - 75 kg 1500 mg > 75 kg 2000 mg Ethambutol < 40 kg 15 mg/kg rounded to nearest 100 mg 40-55 kg 800 mg > 55 kg - 75 kg 1200 mg > 75 kg 1600 mg *For pyrazinamide dosing in patients < 40 kg, 1000 mg used instead of 500 mg
  All treatment is taken daily, for a duration of up to 26 weeks depending on treatment arm.
Period: Per- Protocol
Arm/Group | Regimen 1 - 2EHRZ/4HR (Control Regimen) | Regimen 2 - 2MHRZ/2MHR | Regimen 3 - 2EMRZ/2MR
Started | 640 | 655 | 636
Completed | 510 | 514 | 524
Not Completed | 130 | 141 | 112
Period: Modified Intent to Treat
Arm/Group | Regimen 1 - 2EHRZ/4HR (Control Regimen) | Regimen 2 - 2MHRZ/2MHR | Regimen 3 - 2EMRZ/2MR
Started | 640 | 655 | 636
Completed | 555 | 568 | 551
Not Completed | 85 | 87 | 85

BASELINE CHARACTERISTICS:
Population: Per protocol population
Groups:
- Regimen 2 - 2MHRZ/2MHR (Isoniazid): * Eight weeks of chemotherapy with Moxifloxacin, Isoniazid, Rifampicin and Pyrazinamide plus the Ethambutol placebo, followed by
  * Nine weeks of Moxifloxacin, Isoniazid and Rifampicin, followed by
  * Nine weeks of the Isoniazid placebo and the Rifampicin placebo.
  Moxifloxacin, Ethambutol, Isoniazid, Pyrazinamide & Rifampicin: Moxifloxacin 400 mg Rifampicin < 45 kg 450 mg > 45 kg 600 mg Isoniazid 300 mg Pyrazinamide < 40 kg 25 mg/kg rounded to nearest 500 mg* 40-55 kg 1000 mg > 55 kg - 75 kg 1500 mg > 75 kg 2000 mg Ethambutol < 40 kg 15 mg/kg rounded to nearest 100 mg 40-55 kg 800 mg > 55 kg - 75 kg 1200 mg > 75 kg 1600 mg *For pyrazinamide dosing in patients < 40 kg, 1000 mg used instead of 500 mg
  All treatment is taken daily, for a duration of up to 26 weeks depending on treatment arm.
- Regimen 3 - 2EMRZ/2MR (Ethambutol): * Eight weeks of chemotherapy with Ethambutol, Moxifloxacin, Rifampicin and Pyrazinamide plus the Isoniazid placebo, followed by
  * Nine weeks of Moxifloxacin and Rifampicin plus the Isoniazid placebo, followed by
  * Nine weeks of the Isoniazid placebo and the Rifampicin placebo
  Moxifloxacin, Ethambutol, Isoniazid, Pyrazinamide & Rifampicin: Moxifloxacin 400 mg Rifampicin < 45 kg 450 mg > 45 kg 600 mg Isoniazid 300 mg Pyrazinamide < 40 kg 25 mg/kg rounded to nearest 500 mg* 40-55 kg 1000 mg > 55 kg - 75 kg 1500 mg > 75 kg 2000 mg Ethambutol < 40 kg 15 mg/kg rounded to nearest 100 mg 40-55 kg 800 mg > 55 kg - 75 kg 1200 mg > 75 kg 1600 mg *For pyrazinamide dosing in patients < 40 kg, 1000 mg used instead of 500 mg
  All treatment is taken daily, for a duration of up to 26 weeks depending on treatment arm.
- Total: Total of all reporting groups
Arm/Group | Regimen 1 - 2EHRZ/4HR (Control Regimen) | Regimen 2 - 2MHRZ/2MHR (Isoniazid) | Regimen 3 - 2EMRZ/2MR (Ethambutol) | Total
Number analyzed (Participants) | 510 | 514 | 524 | 1548
Age, Customized [Number; unit: participants]
  < 25 years | 160 | 162 | 146 | 468
  25-35 years | 145 | 162 | 175 | 482
  > 35 years | 205 | 190 | 203 | 598
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 154 | 163 | 155 | 472
  Male | 356 | 351 | 369 | 1076
Race/Ethnicity, Customized [Number; unit: participants]
  Black | 238 | 210 | 237 | 685
  Asian | 160 | 154 | 161 | 475
  Mixed race | 111 | 148 | 126 | 385
  Other | 1 | 2 | 0 | 3
Weight group [Number; unit: participants]
  < 40 kg | 50 | 44 | 58 | 152
  40-45 kg | 80 | 90 | 82 | 252
  > 45-55 kg | 206 | 210 | 204 | 620
  > 55-75 kg | 161 | 158 | 174 | 493
  > 75 kg | 13 | 12 | 6 | 31
Smoking status [Number; unit: participants]
  Never | 246 | 231 | 230 | 707
  Past | 119 | 111 | 134 | 364
  Current | 145 | 172 | 160 | 477
HIV positivity [Number; unit: participants] | 38 | 37 | 35 | 110
Drug resistance [Number; unit: participants]
  Isoniazid | 29 | 34 | 39 | 102
  Pyrazinamide | 14 | 7 | 6 | 27
Cavitation [Number; unit: participants] — Chest cavitation based on blinded assessment of the chest radiograph.
  participants | 368 | 357 | 367 | 1092
Time to positivity on MGIT sputum culture [Number; unit: participants] — Mycobacteria Growth Indicator Tube (MGIT) was used for the detection of mycobacteria.
  participants
    ≥ 5 days | 266 | 263 | 258 | 787
    < 5 days | 229 | 239 | 254 | 722
    Not available | 15 | 12 | 12 | 39

OUTCOME MEASURES:

1. Primary Outcome: Combined Failure of Bacteriological Cure and Relapse Within One Year of Completion of Therapy as Defined by Culture Using Solid Media (Lowenstein-Jensen - LJ).
Description: The primary efficacy outcome was the proportion of patients who had bacteriologically or clinically defined failure or relapse within 18 months after randomization (a composite unfavorable outcome). Culture-negative status was defined as two negative-culture results at different visits without an intervening positive result. The date of culture-negative status was defined as the date of the first negative-culture result. This status continued until there were two positive cultures, without an intervening negative culture, or until there was a single positive culture that was not followed by two negative cultures. Relapse strains were those shown to be identical on 24-locus Mycobacterial interspersed repetitive units (MIRU) analysis. For the final 18 month study visit when both L-J samples were contaminated or missing, if the subject could not be brought back, liquid medium culture results were used in place of solid medium culture results.
Time Frame: 18 months (within one year of completion of therapy)
Population: Per protocol population
Measure: Number; unit: participants with failure or relapse
Arm/Group | Regimen 1 - 2EHRZ/4HR (Control Regimen) | Regimen 2 - 2MHRZ/2MHR | Regimen 3 - 2EMRZ/2MR
Number analyzed (Participants) | 510 | 514 | 524
participants with failure or relapse | 43 | 78 | 105
Statistical Analysis 1: Comparison: Regimen 1 - 2EHRZ/4HR (Control Regimen) vs Regimen 2 - 2MHRZ/2MHR; Test type: Non-Inferiority or Equivalence — Noninferiority was defined as a between-group difference of less than 6 percentage points in the upper boundary of the two-sided 97.5% Wald confidence interval for the difference in proportion of patients with an unfavorable outcome; Adjusted difference in proportions = 6.1, 97.5% CI 2-sided [1.7 to 10.5] — Adjusted difference from control in proportion of unfavorable outcome - percentage points
Statistical Analysis 2: Comparison: Regimen 1 - 2EHRZ/4HR (Control Regimen) vs Regimen 3 - 2EMRZ/2MR; Test type: Non-Inferiority or Equivalence — Noninferiority was defined as a between-group difference of less than 6 percentage points in the upper boundary of the two-sided 97.5% Wald confidence interval for the proportion of patients with an unfavorable outcome; Adjusted difference from control = 11.4, 97.5% CI 2-sided [6.7 to 16.1] — Adjusted difference from control in rate of unfavorable outcome- percentage points

2. Primary Outcome: Number of Patients With Grade 3 or 4 Adverse Events (Using a Modified Division of Acquired Immunodeficiency Syndrome National Institute of Allergy and Infectious Diseases [DAIDS] Scale of Adverse Event Reporting)
Description: The number of participants includes all patients who had at least one grade 3 or 4 adverse event.
Time Frame: 18 months (within one year of completion of therapy)
Population: Safety population, defined as all subjects who underwent randomization and who received at least on dose of study drug.
Measure: Number; unit: participants with Grade 3 or 4 AEs
Arm/Group | Regimen 1 - 2EHRZ/4HR (Control Regimen) | Regimen 2 - 2MHRZ/2MHR | Regimen 3 - 2EMRZ/2MR
Number analyzed (Participants) | 639 | 655 | 636
participants with Grade 3 or 4 AEs | 123 | 127 | 111

3. Secondary Outcome: Combined Failure of Bacteriological Cure and Relapse as Defined by Culture Using Liquid Media (Mycobacteria Growth Indicator Tube-MGIT).
Description: The secondary analysis of efficacy outcome was the proportion of patients who had bacteriologically or clinically defined failure or relapse within 18 months after randomization (a composite unfavorable outcome) based on MGIT. Culture-negative status was defined as two negative-culture results at different visits without an intervening positive result. The date of culture-negative status was defined as the date of the first negative-culture result. This status continued until there were two positive cultures, without an intervening negative culture, or until there was a single positive culture that was not followed by two negative cultures. Relapse strains were those shown to be identical on 24-locus Mycobacterial interspersed repetitive units (MIRU) analysis.
Time Frame: 18 months (within one year of completion of therapy)
Population: Per protocol population
Measure: Number; unit: participants with failure or relapse
Arm/Group | Regimen 1 - 2EHRZ/4HR (Control Regimen) | Regimen 2 - 2MHRZ/2MHR | Regimen 3 - 2EMRZ/2MR
Number analyzed (Participants) | 498 | 498 | 512
participants with failure or relapse | 65 | 98 | 131

4. Secondary Outcome: Number of Patients Who Are Culture Negative (Solid LJ Culture)
Description: Number of patients who are TB LJ culture negative at 8 weeks.
Time Frame: 8 weeks
Population: Per protocol
Measure: Number; unit: participants who are culture negative
Arm/Group | Regimen 1 - 2EHRZ/4HR (Control Regimen) | Regimen 2 - 2MHRZ/2MHR | Regimen 3 - 2EMRZ/2MR
Number analyzed (Participants) | 422 | 457 | 458
participants who are culture negative | 352 | 394 | 401

5. Secondary Outcome: Number of Patients Who Are Culture Negative (Liquid MGIT Culture)
Description: Number of patients who are TB MGIT culture negative at 8 weeks.
Time Frame: 8 weeks
Measure: Number; unit: participants who are culture negative
Arm/Group | Regimen 1 - 2EHRZ/4HR (Control Regimen) | Regimen 2 - 2MHRZ/2MHR | Regimen 3 - 2EMRZ/2MR
Number analyzed (Participants) | 419 | 440 | 429
participants who are culture negative | 235 | 274 | 260

6. Secondary Outcome: Time to First Culture Negative Sputum Sample (LJ Solid Media)
Description: Culture negative for TB using LJ cultures.
Time Frame: 18 months
Population: All randomized patients excluding late screen failures
Measure: Median (95% Confidence Interval); unit: Time to culture negative status / weeks
Arm/Group | Regimen 1 - 2EHRZ/4HR (Control Regimen) | Regimen 2 - 2MHRZ/2MHR | Regimen 3 - 2EMRZ/2MR
Number analyzed (Participants) | 600 | 617 | 604
Time to culture negative status / weeks | 6.0 [6.0 to 6.1] | 6.0 [5.1 to 6] | 6.0 [5.7 to 6.0]

7. Secondary Outcome: Time to First Culture Negative Sputum Sample (MGIT Liquid Media)
Time Frame: 18 months
Population: All randomized patients excluding late screen failures
Measure: Median (95% Confidence Interval); unit: Time to culture negative status / weeks
Arm/Group | Regimen 1 - 2EHRZ/4HR (Control Regimen) | Regimen 2 - 2MHRZ/2MHR | Regimen 3 - 2EMRZ/2MR
Number analyzed (Participants) | 600 | 617 | 604
Time to culture negative status / weeks | 11.9 [8.1 to 12.0] | 8.0 [8.0 to 9.9] | 8.0 [8.0 to 8.1]

8. Secondary Outcome: Sensitivity Analysis Assuming All Losses to Follow-up and Non-tuberculous Deaths Have an Unfavorable Outcome Using Solid (L-J) Media.
Description: Sensitivity Analysis of Primary Efficacy Results of All Randomized Subjects Imputing Unfavorable for Missing Outcomes. Analysis is the number of subjects with an unfavorable outcome. Favorable outcome is defined as the number of subjects with a negative TB culture status at 18 months (at or after 72 weeks), who had not already been classified as having an unfavorable outcome, and whose last positive TB culture result ("isolated positive culture") was followed by at least two negative culture results.
Time Frame: 18 months
Population: All randomized subjects.
Measure: Number; unit: participants with unfavorable outcome
Arm/Group | Regimen 1 - 2EHRZ/4HR (Control Regimen) | Regimen 2 - 2MHRZ/2MHR | Regimen 3 - 2EMRZ/2MR
Number analyzed (Participants) | 640 | 655 | 636
participants with unfavorable outcome | 172 | 219 | 217

9. Secondary Outcome: Sensitivity Analyses Assuming All Losses to Follow-up and Non-tuberculous Deaths Have a Favourable Outcome Using Solid (L-J) Media.
Description: Sensitivity Analysis of Primary Efficacy Results of All Randomized Subjects Imputing Favorable for Missing Outcomes. Analysis is the number of subjects with an unfavorable outcome. Favorable outcome is defined as the number of subjects with a negative TB culture status at 18 months (at or after 72 weeks), who had not already been classified as having an unfavorable outcome, and whose last positive TB culture result ("isolated positive culture") was followed by at least two negative culture results.
Time Frame: 18 months
Measure: Number; unit: participants with unfavorable outcome
Arm/Group | Regimen 1 - 2EHRZ/4HR (Control Regimen) | Regimen 2 - 2MHRZ/2MHR | Regimen 3 - 2EMRZ/2MR
Number analyzed (Participants) | 640 | 655 | 636
participants with unfavorable outcome | 87 | 132 | 132

ADVERSE EVENTS:
Description: Total Number of SAE events and the number and percentage of subjects experiencing each event by system organ class.
Arm/Group | Regimen 1 - 2EHRZ/4HR (Control Regimen) | Regimen 2 - 2MHRZ/2MHR | Regimen 3 - 2EMRZ/2MR
Serious Adverse Events (participants affected / at risk) | 38/639 | 46/655 | 40/636
Other Adverse Events (participants affected / at risk) | 507/639 | 537/655 | 522/636
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regimen 1 - 2EHRZ/4HR (Control Regimen) (N=639) | Regimen 2 - 2MHRZ/2MHR (N=655) | Regimen 3 - 2EMRZ/2MR (N=636)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal Mass (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Abdominal Pain Lower (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0)
Abdominal Tenderness (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Acute Abdomen (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal Disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Peptic Ulcer Perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3) | 6 (11)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea Infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Disseminated Tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Gangrene (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hepatitis B (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Blood Bilirubin Increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood Creatinine Increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Breath Sounds Abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Gamma- Glutamyltransferase Increased (Investigations) | 2 (2) | 0 (0) | 2 (2)
Haemoglobin Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Hepatic Enzyme Increased (Investigations) | 3 (3) | 3 (3) | 4 (4)
International Normalised Ratio Increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Liver Function Test Abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Prothrombin Time prolonged (Investigations) | 0 (0) | 1 (2) | 0 (0)
Respiratory Rate Increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 2 (2) | 6 (8)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 6 (7) | 2 (2)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3) | 0 (0)
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (5) | 3 (3) | 3 (6)
Rales (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 0 (0)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Weight Decreased (Investigations) | 2 (2) | 2 (2) | 2 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regimen 1 - 2EHRZ/4HR (Control Regimen) (N=639) | Regimen 2 - 2MHRZ/2MHR (N=655) | Regimen 3 - 2EMRZ/2MR (N=636)
Abdominal Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 10 (17) | 13 (16) | 8 (11)
Hypochromic Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 8 (13) | 9 (12) | 9 (12)
Lymph Node Pain (Blood and lymphatic system disorders) | 2 (7) | 0 (0) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 1 (2) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 43 (61) | 44 (71) | 50 (68)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Microcytic Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Monocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 4 (13) | 3 (6) | 2 (5)
Neutrophilia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (3)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
Bradycardia (Cardiac disorders) | 2 (3) | 0 (0) | 0 (0)
Cardiac Failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac Failure Congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Congestive Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cor Pulmonale (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperdynamic Left Ventricle (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Left Ventricular Hypertrophy (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 4 (5) | 2 (6)
Pericardial Disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 40 (54) | 48 (71) | 39 (45)
Ventricular Hypertrophy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Auricular Swelling (Ear and labyrinth disorders) | 0 (0) | 1 (2) | 0 (0)
Cerumen Impaction (Ear and labyrinth disorders) | 10 (13) | 5 (7) | 8 (8)
Deafness (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0)
Ear Canal Erythema (Ear and labyrinth disorders) | 2 (2) | 1 (1) | 1 (1)
Ear Discomfort (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 1 (2)
Ear Pain (Ear and labyrinth disorders) | 1 (1) | 3 (4) | 5 (7)
Ear Pruritus (Ear and labyrinth disorders) | 2 (2) | 1 (1) | 0 (0)
Haematotympanum (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Hearing Impaired (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (2)
Otorrhoea (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1)
Tympanic Membrane Hyperaemia (Ear and labyrinth disorders) | 0 (0) | 4 (4) | 1 (1)
Tympanic Membrane Perforation (Ear and labyrinth disorders) | 2 (4) | 4 (4) | 3 (4)
Tympanic Membrane Scarring (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Tympanosclerosis (Ear and labyrinth disorders) | 1 (2) | 4 (6) | 1 (2)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 3 (3) | 0 (0)
Astigmatism (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 2 (2) | 0 (0) | 4 (4)
Conjunctival Haemorrhage (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Conjunctival Hyperaemia (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Conjunctival Irritation (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Conjunctival Pallor (Eye disorders) | 1 (1) | 3 (3) | 3 (3)
Conjunctivitis (Eye disorders) | 2 (2) | 4 (6) | 3 (3)
Conjunctivitis Allergic (Eye disorders) | 3 (3) | 2 (2) | 3 (3)
Corneal Opacity (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Dry Eye (Eye disorders) | 1 (1) | 2 (2) | 0 (0)
Eye Irritation (Eye disorders) | 0 (0) | 2 (2) | 2 (2)
Eye Oedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eye Pain (Eye disorders) | 4 (4) | 2 (2) | 4 (4)
Eye Pruritus (Eye disorders) | 4 (4) | 5 (6) | 8 (9)
Eyelid Oedema (Eye disorders) | 2 (2) | 0 (0) | 1 (1)
Eyelids Pruritus (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Hypermetropia (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Keratitis (Eye disorders) | 1 (1) | 0 (0) | 1 (2)
Lacrimation Increased (Eye disorders) | 2 (2) | 1 (1) | 2 (2)
Night Blindness (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Ocular Discomfort (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Ocular Hyperaemia (Eye disorders) | 1 (1) | 0 (0) | 2 (3)
Ocular Icterus (Eye disorders) | 2 (2) | 2 (2) | 1 (1)
Photophobia (Eye disorders) | 2 (2) | 2 (2) | 1 (1)
Pterygium (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Scleral Hyperaemia (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Scleritis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Uveitis (Eye disorders) | 0 (0) | 1 (3) | 0 (0)
Vision Blurred (Eye disorders) | 10 (12) | 8 (8) | 9 (9)
Visual Acuity Reduced (Eye disorders) | 7 (9) | 16 (18) | 12 (12)
Visual Impairment (Eye disorders) | 4 (5) | 3 (3) | 1 (2)
Vitreous Floaters (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal Discomfort (Gastrointestinal disorders) | 1 (1) | 5 (6) | 7 (8)
Abdominal Distension (Gastrointestinal disorders) | 3 (3) | 2 (3) | 4 (4)
Abdominal Pain (Gastrointestinal disorders) | 12 (17) | 15 (20) | 15 (17)
Abdominal Pain Lower (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 10 (10) | 14 (14) | 7 (8)
Abdominal Rigidity (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal Tenderness (Gastrointestinal disorders) | 5 (5) | 9 (13) | 6 (8)
Anal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Anal Pruritus (Gastrointestinal disorders) | 1 (2) | 2 (3) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0)
Chapped Lips (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 10 (11) | 12 (17) | 3 (3)
Dental Caries (Gastrointestinal disorders) | 6 (6) | 1 (1) | 7 (9)
Diarrhoea (Gastrointestinal disorders) | 16 (18) | 38 (51) | 46 (59)
Dyspepsia (Gastrointestinal disorders) | 10 (13) | 8 (8) | 5 (6)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Epigastric Discomfort (Gastrointestinal disorders) | 3 (3) | 1 (1) | 2 (2)
Faecal Volume Increased (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0)
Food Poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Frequent Bowel Movements (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 4 (5) | 7 (7) | 3 (4)
Gastrointestinal Hypermotility (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal Pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Gastrointestinal Sounds Abnormal (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1)
Gingival Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gingival Recession (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Glossitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (3)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 3 (4) | 1 (1) | 3 (3)
Hyperchlorhydria (Gastrointestinal disorders) | 3 (3) | 3 (3) | 0 (0)
Lip Blister (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lip Swelling (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Lip Ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Mouth Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 40 (49) | 39 (44) | 45 (50)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (3)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oral Mucosal Discolouration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Oral Pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Paraesthesia Oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Parotid Gland Enlargement (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Peptic Ulcer (Gastrointestinal disorders) | 2 (3) | 2 (3) | 0 (0)
Post-Tussive Vomiting (Gastrointestinal disorders) | 1 (1) | 4 (5) | 1 (2)
Rectal Discharge (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rectal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal Tenesmus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Salivary Gland Disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Salivary Gland Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Tongue Coated (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Tongue Disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Tongue Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Tongue Ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 5 (7) | 5 (6) | 4 (4)
Vomiting (Gastrointestinal disorders) | 44 (56) | 70 (95) | 70 (92)
Adhesion (General disorders) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 12 (14) | 10 (11) | 16 (19)
Catheter Site Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Chest Discomfort (General disorders) | 2 (2) | 4 (4) | 1 (1)
Chest Pain (General disorders) | 60 (76) | 49 (57) | 55 (68)
Chills (General disorders) | 3 (3) | 1 (2) | 0 (0)
Crepitations (General disorders) | 5 (5) | 4 (4) | 7 (8)
Face Oedema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 10 (12) | 21 (22) | 7 (7)
Gait Disturbance (General disorders) | 0 (0) | 1 (1) | 0 (0)
Generalised Oedema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hernia (General disorders) | 1 (1) | 0 (0) | 1 (1)
Hypothermia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Influenza Like Illness (General disorders) | 2 (2) | 0 (0) | 0 (0)
Local Swelling (General disorders) | 5 (7) | 9 (10) | 2 (2)
Malaise (General disorders) | 2 (2) | 3 (3) | 3 (3)
Mass (General disorders) | 0 (0) | 1 (1) | 0 (0)
Medical Device Pain (General disorders) | 0 (0) | 1 (1) | 1 (1)
Mucosal Discolouration (General disorders) | 0 (0) | 2 (2) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 20 (22) | 18 (20) | 23 (30)
Oedema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Oedema Peripheral (General disorders) | 6 (7) | 2 (3) | 2 (4)
Pain (General disorders) | 10 (12) | 9 (14) | 10 (17)
Pyrexia (General disorders) | 58 (95) | 67 (103) | 84 (116)
Tenderness (General disorders) | 0 (0) | 0 (0) | 1 (1)
Thirst (General disorders) | 1 (1) | 1 (1) | 0 (0)
Unevaluable Event (General disorders) | 0 (0) | 0 (0) | 1 (1)
Xerosis (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic Function Abnormal (Hepatobiliary disorders) | 5 (10) | 2 (3) | 2 (2)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (3)
Hepatomegaly (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 (3) | 5 (7) | 2 (3)
Jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Liver Tenderness (Hepatobiliary disorders) | 0 (0) | 2 (2) | 1 (2)
Abscess Neck (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Acarodermatitis (Infections and infestations) | 2 (3) | 1 (2) | 1 (1)
Amoebic Dysentery (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Anal Abscess (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Body Tinea (Infections and infestations) | 1 (1) | 5 (5) | 3 (4)
Breast Abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Bronchitis (Infections and infestations) | 10 (10) | 3 (3) | 6 (6)
Bronchitis Bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchitis Viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Candida Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Chest Wall Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Dermatitis Infected (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Dysentery (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Ear Infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Eye Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Febrile Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Fungal Infection (Infections and infestations) | 2 (3) | 2 (2) | 2 (2)
Fungal Skin Infection (Infections and infestations) | 5 (7) | 3 (3) | 3 (5)
Furuncle (Infections and infestations) | 1 (2) | 0 (0) | 2 (3)
Gastroenteritis (Infections and infestations) | 5 (6) | 1 (1) | 13 (14)
Gastroenteritis Viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Genital Candidiasis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Genital Herpes (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Giardiasis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Gingival Abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Helminthic Infection (Infections and infestations) | 1 (2) | 2 (2) | 2 (2)
Herpes Zoster (Infections and infestations) | 2 (2) | 4 (5) | 1 (1)
Hiv Infection (Infections and infestations) | 2 (3) | 1 (1) | 0 (0)
Impetigo (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Infected Dermal Cyst (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infected Skin Ulcer (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 15 (16) | 16 (16) | 17 (22)
Laryngitis (Infections and infestations) | 3 (3) | 1 (1) | 3 (3)
Lobar Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 3 (3)
Lower Respiratory Tract Infection (Infections and infestations) | 5 (5) | 10 (11) | 4 (4)
Lower Respiratory Tract Infection Bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Lung Abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lung Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Malaria (Infections and infestations) | 15 (15) | 10 (11) | 9 (10)
Molluscum Contagiosum (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Mycobacterium Fortuitum Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Myringitis (Infections and infestations) | 1 (3) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 12 (14) | 15 (16) | 20 (21)
Oesophageal Candidiasis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Onychomycosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Ophthalmic Herpes Zoster (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Oral Candidiasis (Infections and infestations) | 6 (9) | 12 (14) | 11 (13)
Oral Hairy Leukoplakia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Oral Herpes (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Otitis Externa (Infections and infestations) | 0 (0) | 2 (3) | 0 (0)
Otitis Media (Infections and infestations) | 2 (2) | 2 (3) | 0 (0)
Otitis Media Chronic (Infections and infestations) | 1 (2) | 1 (1) | 0 (0)
Pelvic Inflammatory Disease (Infections and infestations) | 1 (1) | 1 (2) | 1 (1)
Pericarditis Tuberculous (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 3 (3) | 7 (8) | 7 (7)
Pharyngotonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumocystis Jirovecii Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 6 (9) | 3 (5) | 7 (7)
Pneumonia Bacterial (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pneumonia Haemophilus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pulmonary Tuberculosis (Infections and infestations) | 14 (14) | 24 (27) | 36 (37)
Pulpitis Dental (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Rash Pustular (Infections and infestations) | 0 (0) | 1 (1) | 2 (4)
Respiratory Tract Infection (Infections and infestations) | 1 (1) | 2 (3) | 3 (3)
Respiratory Tract Infection Viral (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 10 (11) | 13 (16) | 18 (21)
Schistosomiasis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Schistosomiasis Bladder (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Septic Rash (Infections and infestations) | 0 (0) | 0 (0) | 1 (8)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (3)
Subcutaneous Abscess (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Tinea Capitis (Infections and infestations) | 1 (1) | 4 (5) | 0 (0)
Tinea Faciei (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tinea Infection (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Tinea Pedis (Infections and infestations) | 2 (2) | 0 (0) | 3 (4)
Tinea Versicolour (Infections and infestations) | 1 (1) | 3 (3) | 4 (5)
Tonsillitis (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Tooth Abscess (Infections and infestations) | 1 (2) | 2 (2) | 1 (2)
Tooth Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tuberculosis (Infections and infestations) | 3 (3) | 11 (11) | 8 (9)
Tuberculosis Gastrointestinal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Typhoid Fever (Infections and infestations) | 3 (3) | 0 (0) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 24 (27) | 20 (23) | 20 (24)
Upper Respiratory Tract Infection Bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 8 (9) | 7 (8) | 11 (12)
Vaginitis Bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Varicella (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Viral Infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 7 (13) | 6 (11) | 7 (11)
Vulvovaginal Candidiasis (Infections and infestations) | 5 (8) | 7 (9) | 6 (8)
Vulvovaginitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Wound Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Wound Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Accident (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Animal Bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Ankle Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 4 (4)
Excoriation (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 2 (2)
Eyelid Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fibula Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Foreign Body (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Foreign Body In Eye (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hand Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Human Bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Humerus Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Incorrect Dose Administered (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Injury Corneal (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Jaw Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Joint Injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (3) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 4 (5)
Ligament Sprain (Injury, poisoning and procedural complications) | 0 (0) | 2 (4) | 2 (2)
Lip Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2)
Muscle Strain (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 1 (1)
Periorbital Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Rib Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Scar (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0)
Skeletal Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Soft Tissue Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 3 (3)
Stab Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Subdural Haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Thermal Burn (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 1 (1)
Tibia Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tooth Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1)
Activated Partial Thromboplastin Time Prolonged (Investigations) | 10 (13) | 10 (13) | 13 (16)
Alanine Aminotransferase Abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Alanine Aminotransferase Decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 25 (37) | 30 (39) | 16 (24)
Amylase Increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 28 (41) | 35 (47) | 24 (31)
Blood Albumin Decreased (Investigations) | 1 (3) | 2 (3) | 2 (2)
Blood Bilirubin Increased (Investigations) | 4 (4) | 9 (14) | 2 (6)
Blood Creatine Increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Blood Creatinine Decreased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Blood Creatinine Increased (Investigations) | 7 (8) | 15 (17) | 7 (10)
Blood Glucose Abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood Glucose Increased (Investigations) | 2 (4) | 3 (9) | 0 (0)
Blood Potassium Decreased (Investigations) | 0 (0) | 3 (3) | 4 (5)
Blood Potassium Increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Blood Pressure Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood Pressure Diastolic Decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood Pressure Diastolic Increased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Blood Pressure Increased (Investigations) | 6 (7) | 6 (7) | 7 (8)
Blood Pressure Systolic Decreased (Investigations) | 0 (0) | 1 (1) | 2 (2)
Blood Pressure Systolic Increased (Investigations) | 2 (2) | 1 (4) | 0 (0)
Blood Sodium Decreased (Investigations) | 4 (9) | 2 (2) | 0 (0)
Blood Sodium Increased (Investigations) | 0 (0) | 0 (0) | 4 (5)
Blood Urea Increased (Investigations) | 1 (1) | 1 (2) | 0 (0)
Blood Uric Acid Increased (Investigations) | 2 (2) | 1 (1) | 0 (0)
Body Temperature Increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Breath Sounds Abnormal (Investigations) | 7 (9) | 9 (10) | 5 (6)
Cardiac Murmur (Investigations) | 0 (0) | 0 (0) | 1 (1)
Cd4 Lymphocytes Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Chest X-Ray Abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Coagulation Test Abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Colour Vision Tests Abnormal (Investigations) | 0 (0) | 1 (2) | 0 (0)
Creatinine Renal Clearance Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Gamma-Glutamyltransferase Increased (Investigations) | 2 (4) | 1 (1) | 0 (0)
Gastrointestinal Examination Abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Glucose Urine Present (Investigations) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin Decreased (Investigations) | 13 (24) | 18 (29) | 20 (28)
Heart Rate Increased (Investigations) | 2 (2) | 0 (0) | 1 (1)
Heart Rate Irregular (Investigations) | 3 (3) | 1 (1) | 1 (3)
Heart Sounds Abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hepatic Enzyme Abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hepatic Enzyme Increased (Investigations) | 22 (36) | 18 (30) | 11 (17)
International Normalised Ratio Abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
International Normalised Ratio Increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Liver Function Test Abnormal (Investigations) | 2 (4) | 0 (0) | 0 (0)
Liver Palpable Subcostal (Investigations) | 0 (0) | 0 (0) | 1 (2)
Lymph Node Palpable (Investigations) | 0 (0) | 0 (0) | 2 (2)
Neutrophil Count Decreased (Investigations) | 1 (1) | 3 (3) | 0 (0)
Neutrophil Percentage Decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Ophthalmological Examination Abnormal (Investigations) | 0 (0) | 1 (2) | 0 (0)
Percussion Test Abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Platelet Count Decreased (Investigations) | 5 (5) | 3 (6) | 4 (4)
Prothrombin Level Increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Prothrombin Time Abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
Prothrombin Time Prolonged (Investigations) | 11 (15) | 13 (16) | 20 (30)
Pulmonary Physical Examination Abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
Red Blood Cell Sedimentation Rate Increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Respiratory Rate Increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Transaminases Increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Urine Analysis Abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Urine Cytology Abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
Urine Leukocyte Esterase Positive (Investigations) | 1 (1) | 0 (0) | 0 (0)
Weight Decreased (Investigations) | 62 (83) | 70 (85) | 72 (77)
White Blood Cell Count Decreased (Investigations) | 2 (3) | 0 (0) | 1 (2)
White Blood Cell Count Increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Abnormal Loss Of Weight (Metabolism and nutrition disorders) | 15 (22) | 20 (23) | 16 (18)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 45 (54) | 33 (35) | 45 (50)
Dehydration (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 1 (1)
Diabetes Mellitus (Metabolism and nutrition disorders) | 6 (10) | 7 (9) | 9 (13)
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 1 (1)
Electrolyte Imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3) | 3 (6) | 2 (5)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 3 (3)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (3) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (4) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (5) | 5 (6) | 1 (1)
Iron Deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Metabolic Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Polydipsia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Vitamin B Complex Deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (182) | 12 (177) | 10 (162)
Arthritis (Musculoskeletal and connective tissue disorders) | 6 (7) | 6 (12) | 1 (1)
Arthropathy (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (7) | 2 (2)
Arthrotoxicity (Musculoskeletal and connective tissue disorders) | 1 (2) | 3 (5) | 4 (7)
Back Pain (Musculoskeletal and connective tissue disorders) | 19 (26) | 20 (24) | 20 (22)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 1 (1)
Chondrotoxicity (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 1 (1)
Clubbing (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (3) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Finger Deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 4 (4)
Gouty Arthritis (Musculoskeletal and connective tissue disorders) | 2 (4) | 0 (0) | 1 (1)
Joint Range Of Motion Decreased (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 1 (1)
Joint Stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3) | 1 (1)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 5 (6) | 4 (5) | 6 (9)
Ligament Pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (3) | 0 (0)
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 0 (0)
Muscle Atrophy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle Fatigue (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 10 (11) | 6 (10) | 4 (4)
Muscle Swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 3 (4) | 5 (5) | 2 (2)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (5) | 0 (0)
Musculoskeletal Discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal Disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 12 (17) | 11 (12) | 7 (8)
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 4 (5) | 4 (6) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 14 (15) | 28 (41) | 21 (25)
Myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Neck Pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 6 (6) | 2 (3)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 32 (44) | 27 (38) | 29 (43)
Periarthritis (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0) | 0 (0)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3) | 0 (0)
Sensation Of Heaviness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal Pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Synovial Cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Tendon Disorder (Musculoskeletal and connective tissue disorders) | 2 (3) | 5 (6) | 4 (4)
Tendon Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4) | 3 (3)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3) | 1 (1)
Trigger Finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Upper Extremity Mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Anogenital Warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Penile Wart (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Pharyngeal Neoplasm Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Thyroid Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Ageusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Burning Sensation (Nervous system disorders) | 2 (3) | 3 (3) | 0 (0)
Coma (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 15 (17) | 16 (25) | 26 (32)
Dizziness Postural (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 35 (44) | 39 (45) | 52 (63)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hemiplegia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperreflexia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 8 (14) | 8 (9) | 12 (19)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3)
Loss Of Consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Memory Impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Neuritis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Neuropathy Peripheral (Nervous system disorders) | 13 (16) | 6 (6) | 11 (14)
Paraesthesia (Nervous system disorders) | 8 (12) | 10 (13) | 3 (5)
Parosmia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Post Herpetic Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Restless Legs Syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 2 (3)
Sensory Disturbance (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 6 (6) | 5 (8) | 7 (7)
Syncope (Nervous system disorders) | 2 (2) | 1 (1) | 2 (2)
Tension Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Visual Field Defect (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Abortion Threatened (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 4 (4) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 2 (2) | 5 (5)
Anxiety Disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Confusional State (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (3)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Initial Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 12 (16) | 6 (6) | 6 (6)
Nervousness (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Premature Ejaculation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Psychotic Disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Sleep Disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Tension (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Bilirubinuria (Renal and urinary disorders) | 0 (0) | 5 (5) | 0 (0)
Dysuria (Renal and urinary disorders) | 6 (7) | 5 (5) | 2 (2)
Enuresis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Glycosuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 3 (5)
Haematuria (Renal and urinary disorders) | 2 (2) | 3 (3) | 4 (6)
Leukocyturia (Renal and urinary disorders) | 1 (1) | 4 (4) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (2) | 0 (0) | 1 (1)
Polyuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 3 (3) | 6 (6) | 7 (8)
Renal Colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2)
Renal Failure Acute (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Urethral Discharge (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary Incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Breast Discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Breast Pain (Reproductive system and breast disorders) | 2 (4) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 1 (1)
Erectile Dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Fibrocystic Breast Disease (Reproductive system and breast disorders) | 1 (2) | 0 (0) | 0 (0)
Genital Rash (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (2)
Genital Ulceration (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Menometrorrhagia (Reproductive system and breast disorders) | 1 (4) | 0 (0) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Menstruation Irregular (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0)
Nipple Pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Penile Discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Polymenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus Genital (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1)
Testicular Pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Vaginal Discharge (Reproductive system and breast disorders) | 1 (1) | 2 (2) | 1 (1)
Vaginal Disorder (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Vaginal Haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal Pruritus (Reproductive system and breast disorders) | 1 (1) | 4 (4) | 1 (1)
Allergic Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 5 (7) | 4 (4)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 85 (107) | 11 (136) | 13 (188)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 49 (70) | 54 (67) | 79 (99)
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) | 2 (3)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 51 (59) | 55 (71) | 40 (47)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 5 (8) | 8 (9) | 5 (6)
Mediastinal Shift (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0)
Nasal Discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 0 (0)
Nasal Obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
Nasal Oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Nasal Ulcer (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Obstructive Airways Disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 10 (10) | 11 (11)
Pharyngeal Erythema (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 4 (4)
Pharyngeal Oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (3)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pleural Rub (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 5 (6) | 18 (19)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (4) | 10 (10)
Pulmonary Arterial Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (2) | 1 (1)
Pulmonary Hilum Mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rales (Respiratory, thoracic and mediastinal disorders) | 11 (17) | 10 (11) | 18 (20)
Respiratory Disorder (Respiratory, thoracic and mediastinal disorders) | 46 (58) | 52 (63) | 54 (69)
Respiratory Fremitus (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (4) | 5 (5)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 11 (12) | 7 (8) | 4 (5)
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (5) | 2 (2)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0)
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Tonsillar Hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Tonsillar Inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Upper-Airway Cough Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 6 (10) | 7 (8) | 9 (11)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 4 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Chloasma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dermal Cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 6 (7) | 4 (5) | 3 (3)
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 1 (1)
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 2 (2)
Dermatitis Bullous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (1) | 0 (0)
Diabetic Foot (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dry Skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (3)
Exfoliative Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Hand Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Intertrigo (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Milia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Night Sweats (Skin and subcutaneous tissue disorders) | 29 (32) | 48 (50) | 57 (61)
Pemphigus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 39 (46) | 35 (52) | 37 (47)
Pruritus Generalised (Skin and subcutaneous tissue disorders) | 18 (22) | 16 (20) | 9 (12)
Rash (Skin and subcutaneous tissue disorders) | 25 (33) | 18 (20) | 22 (32)
Rash Generalised (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 0 (0)
Rash Macular (Skin and subcutaneous tissue disorders) | 4 (5) | 5 (7) | 2 (2)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 5 (6) | 4 (4) | 4 (4)
Rash Maculovesicular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash Papular (Skin and subcutaneous tissue disorders) | 6 (6) | 7 (8) | 8 (13)
Rash Pruritic (Skin and subcutaneous tissue disorders) | 9 (12) | 4 (4) | 5 (8)
Seborrhoeic Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Skin Discolouration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0)
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 1 (1)
Skin Hypopigmentation (Skin and subcutaneous tissue disorders) | 2 (4) | 2 (2) | 0 (0)
Skin Lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (3)
Skin Reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 1 (1)
Skin Warm (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Swelling Face (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 0 (0)
Cosmetic Body Piercing (Social circumstances) | 1 (1) | 0 (0) | 0 (0)
Physical Assault (Social circumstances) | 3 (3) | 0 (0) | 0 (0)
Victim Of Crime (Social circumstances) | 2 (2) | 1 (1) | 2 (2)
Cataract Operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Ear Operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Eye Prosthesis Insertion (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Finger Amputation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Leg Amputation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Tooth Extraction (Surgical and medical procedures) | 2 (2) | 2 (2) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 1 (3) | 0 (0) | 1 (1)
Diastolic Hypertension (Vascular disorders) | 1 (2) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hot Flush (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 15 (28) | 18 (30) | 10 (16)
Hypertensive Crisis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 1 (1) | 5 (5)
Orthostatic Hypotension (Vascular disorders) | 2 (2) | 0 (0) | 2 (2)
Pallor (Vascular disorders) | 2 (2) | 4 (4) | 1 (1)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Poor Peripheral Circulation (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Systolic Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Varicose Vein (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No